CLINICAL TRIAL: NCT01217346
Title: A Prevalence Study of Obstructive Sleep Apnea in Subjects With Chest Pain, Positive Exercise Treadmill Test and Normal Coronary Angiogram
Status: Terminated | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Lui Mei Sze Macy, Queen Mary Hospital, The University of Hong Kong
Other Study IDs: UW 09-127
Record Dates: First submitted 2010-10-04; First posted 2010-10-08 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Obstructive Sleep Apnea; Cardiac Syndrome X; Endothelial Dysfunction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microvascular Angina

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cardiac syndrome X: subjects fulfilling the clinical triad of cardiac syndrome X
  Interventions: Other: no intervention is involved in this study

INTERVENTIONS:
Other: no intervention is involved in this study — no intervention is involved in this study

SUMMARY:
Cardiac syndrome X consists of a triad of chest pain, abnormal exercise stress testing and normal coronary angiogram, and is hypothesized to be related to endothelial dysfunction. Endothelial dysfunction is also reported to be linked to obstructive sleep apnea. While chest pain can be one of potential presenting symptoms of obstructive sleep apnea, the investigators hypothesize that obstructive sleep apnea is common in subjects with cardiac syndrome X.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧18 years, < 70 years
* Symptom of chest pain occurring at least once in the preceding year
* Positive exercise treadmill test
* Negative coronary angiogram
* Mentally fit to give informed consent

Exclusion Criteria:

* Mentally incapacitated persons
* Congestive heart failure
* Other potential causes of orthopnea (severe chronic obstructive pulmonary disease, persistent asthma)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chest pain, positive exercise treadmill test and normal coronary angiogram
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
apnea hypopnea index | measure at a single time point when the subjects are admitted for overnight polysomnography
  assess apnea hypopnea index by overnight polysomnography, by a single admission to sleep laboratory

SECONDARY OUTCOMES:
endothelial function | measured at a single time point when the subjects are admitted for overnight polysomnography
  assess endothelial function by EndoPAT 2000 (an non-invasive device) and peripheral blood endothelial progenitor cells

CONTACTS AND LOCATIONS:
Overall Officials: Macy MS Lui, Principal Investigator — Queen Mary Hospital, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Ip MS, Tse HF, Lam B, Tsang KW, Lam WK. Endothelial function in obstructive sleep apnea and response to treatment. Am J Respir Crit Care Med. 2004 Feb 1;169(3):348-53. doi: 10.1164/rccm.200306-767OC. Epub 2003 Oct 9. PMID 14551167
- [Background] Loui WS, Blackshear JL, Fredrickson PA, Kaplan J. Obstructive sleep apnea manifesting as suspected angina: report of three cases. Mayo Clin Proc. 1994 Mar;69(3):244-8. doi: 10.1016/s0025-6196(12)61063-5. PMID 8133662
- [Background] Philip P, Guilleminault C. ST segment abnormality, angina during sleep and obstructive sleep apnea. Sleep. 1993 Sep;16(6):558-9. doi: 10.1093/sleep/16.6.558. No abstract available. PMID 8235241
- [Background] Chan HS, Chiu HF, Tse LK, Woo KS. Obstructive sleep apnea presenting with nocturnal angina, heart failure, and near-miss sudden death. Chest. 1991 Apr;99(4):1023-5. doi: 10.1378/chest.99.4.1023. PMID 2009755
- [Background] Melikian N, De Bruyne B, Fearon WF, MacCarthy PA. The pathophysiology and clinical course of the normal coronary angina syndrome (cardiac syndrome X). Prog Cardiovasc Dis. 2008 Jan-Feb;50(4):294-310. doi: 10.1016/j.pcad.2007.01.003. No abstract available. PMID 18156008